CLINICAL TRIAL: NCT04973865
Title: Cross Cultural Adaptation of International Physical Activity Questionaire Short Form in Urdu Version
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC00758 Syeda Sumaira
Record Dates: First submitted 2021-07-17; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Heart Diseases
Keywords: IPAQ-SF; 6MWT; Rate pressure product
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Population: 50 Patients who have chronic diseases, such as cardiovascular, will consider as high risk, those who have more than two number of CAD risk factor will categorize as mild and patients have less than two risk factor of CAD will consider as low risk factor. (ACSM risk stratification guide lines)
  Interventions: Other: Validation & reliability
- Healthy: 30 Healthy individual with no cardiac diseased.
  Interventions: Other: Validation & reliability

INTERVENTIONS:
Other: Validation & reliability — Translated version of IPAQ(SF) validation & Reliability
  Other Names: Translated Tool

SUMMARY:
The IPAQ-SF scale is widely used in our clinical settings. The translated version of IPAQ-SF scale in Urdu will help the clinician in collecting data thus, easy to understand for the patient and making it more desirable in our region.

DETAILED DESCRIPTION:
The purpose of study is to translate IPAQ-SF (International Physical Activity Questionnaire- short form) scale in Urdu and to determine the validity & reliability of IPAQ-SF in Urdu version. Patients who are at high risk of chronic diseases such as cardiovascular disease, diabetes, and hypertension age between 30 to 65 years and can understand Urdu and English language are included in my study. 6mint walk test performed to assess aerobic capacity and endurance and physical activity over the last seven days is recorded on the translated version of IPAQ-SF in Urdu and then back of Urdu into English.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic diseases, such as cardiovascular, pulmonary and metabolic disease will consider as high risk, those who have more than two number of CAD risk factor will categorize as mild and patients have less than two risk factor of CAD will consider as low risk factor.(ACSM risk stratification guide lines)

Those who can read and understand English and Urdu as well.

Exclusion Criteria:

* Those with known Parkinson's disease, cerebrovascular disease or dementia.

Individuals have difficulty with reading because of low educational level

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diseased and Healthy individual group to evaluate the Physical Activity and do validation of IPAQ Short form Urdu Version. Test retest reliability in both group for IPQ short form urdu version.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Rate Pressure Product | One day
  Rate pressure product is amount of stress on cardiac muscle during each beat and amount of blood pressure exert against arterial circulation (SBP).
6 minute Walk Test | One day
  Area that is covered during six minutes shows the result with whom functional capability is compared. Walkway with no obstruction and an area of thirty meter is used and patient is told to keep walking for the duration of six minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MS, Principal Investigator — Riphah International University; Iqbal Tariq, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hervas G, Ruiz-Litago F, Irazusta J, Fernandez-Atutxa A, Fraile-Bermudez AB, Zarrazquin I. Physical Activity, Physical Fitness, Body Composition, and Nutrition Are Associated with Bone Status in University Students. Nutrients. 2018 Jan 10;10(1):61. doi: 10.3390/nu10010061. PMID 29320446
- [Background] Helou K, El Helou N, Mahfouz M, Mahfouz Y, Salameh P, Harmouche-Karaki M. Validity and reliability of an adapted arabic version of the long international physical activity questionnaire. BMC Public Health. 2017 Jul 24;18(1):49. doi: 10.1186/s12889-017-4599-7. PMID 28738790
- [Background] Macfarlane DJ, Lee CC, Ho EY, Chan KL, Chan DT. Reliability and validity of the Chinese version of IPAQ (short, last 7 days). J Sci Med Sport. 2007 Feb;10(1):45-51. doi: 10.1016/j.jsams.2006.05.003. Epub 2006 Jun 30. PMID 16807105